CLINICAL TRIAL: NCT01598428
Title: Effect of Anterior Capsule Polishing on Effective Lens Position After Cataract Surgery
Brief Title: Anterior Capsule Polishing Effect on Effective Lens Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yang Gao, Principal Investigator, Shandong University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: YGao
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Cataract
Keywords: age related cataract; phacoemulsification; anterior capsule polishing; optical coherence tomography; anterior chamber depth
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- cataract (Other)
  Interventions: Procedure: anterior capsule polishing

INTERVENTIONS:
Procedure: anterior capsule polishing — polish the anterior capsule and the equator of capsule extensively with a Whitman Shepherd Double-Ended Capsule Polisher

SUMMARY:
* The purpose of this study is to evaluate effects of anterior capsule polishing on effective lens position (ELP) and actual axial movement of the intraocular lens (IOL) by measuring anterior chamber depth (ACD)
* patients with bilateral age-related cataract undergo bilateral uneventful cataract surgeries with in-the- bag implantation of a single-piece hydrophobic acrylic foldable IOL (SN60WF). The anterior capsule was extensively polished using Whitman Shepherd Double-Ended Capsule Polisher in one eye randomly, and the other not. The ACD was measured 1day, 1 week, 1month, 3 months and 6 months with anterior segment Optical Coherence Tomograph (AS-OCT) postoperatively. The actual axial movement of IOL was defined as the root mean square (RMS) of the change in ELP at each visit.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* good overall physical constitution
* uneventful surgeries of both eyes with in-the-bag IOL implantation

Exclusion Criteria:

* history of intraocular surgery or laser therapy
* history of ocular trauma or ocular disease
* high myopia
* diabetes
* severe retinal pathology
* patients who could not return on time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophtalmology,Qianfoshan Hospital,Shandong University, Jinan, Shandong, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Cataract: During cataract surgery, the anterior capsule was unpolished intraoperatively in one eye; the anterior capsule and the equator of capsule was extensively polished intraoperatively in the other eye. Anterior capsule polishing: polish the anterior capsule and the equator of capsule extensively with a Whitman Shepherd Double-Ended Capsule Polisher
Period: Overall Study
Arm/Group | Cataract
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cataract
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  China | 20

OUTCOME MEASURES:

1. Primary Outcome: Effective Lens Position
Description: Effective lens position was measured with anterior chamber depth 1 day，1 week, 1 month as well as 3 months and 6 months postoperatively using anterior segment Optical Coherence Tomograph. The anterior chamber depth defined as the distance between the posterior surface of the corneal and anterior surface of intraocular lens in the pupil center along the optical axis. The actual movement of intraocular lenses was defined as the root mean square of changes in the effective lens position at each visit.
Time Frame: 1 day，1 week, 1 month，3 months and 6 months postoperatively
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Groups:
- Control: During cataract surgery, the anterior capsule was unpolished intraoperatively in this eye;
- Anterior Capsule Polishing: During cataract surgery, the anterior capsule and the equator of capsule was extensively polished intraoperatively in this eye. Anterior capsule polishing: polish the anterior capsule and the equator of capsule extensively with a Whitman Shepherd Double-Ended Capsule Polisher
Arm/Group | Control | Anterior Capsule Polishing
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
mm
  ELP 1 day postoperative | 3.97 (0.27) | 4.02 (0.32)
  ELP 1 week postoperative | 3.93 (0.25) | 3.99 (0.29)
  ELP 1 month postoperative | 3.97 (0.23) | 3.99 (0.26)
  ELP 3 months postoperative | 3.98 (0.24) | 3.97 (0.27)
  ELP 6 months postoperative | 3.92 (0.25) | 3.97 (0.28)
  the root mean square of changes in the ELP(ELPrms) | 0.06 (0.02) | 0.05 (0.02)

2. Secondary Outcome: Uncorrected Visual Acuity(UCVA)
Description: The UCVA was recorded in logMAR units at each vist
Time Frame: 1 day，1 week, 1 month as well as 3 months and 6 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Control | Anterior Capsule Polishing
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
logMAR
  UCVA 1 day postoperative | 0.07 (0.10) | 0.07 (0.09)
  UCVA 1 week postoperative | 0.08 (0.09) | 0.08 (0.09)
  UCVA 1 month postoperative | 0.09 (0.10) | 0.08 (0.09)
  UCVA 3 months postoperative | 0.10 (0.12) | 0.10 (0.08)
  UCVA 6 months postoperative | 0.10 (0.11) | 0.10 (0.08)

3. Secondary Outcome: Refractive Error
Description: auto refraction was performed at each visit. Spherical equivalent refraction (SER) (sphere +cylinder/2) was used in subsequent calculations.
Time Frame: 1 day，1 week, 1 month as well as 3 months and 6 months postoperatively
Measure: Mean (Standard Deviation); unit: diopter(D)
Units Other Than Participants: eyes
Arm/Group | Control | Anterior Capsule Polishing
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
diopter(D)
  the refractive error 1 day postoperative | -0.33 (0.18) | -0.45 (0.18)
  the refractive error 1 week postoperative | -0.42 (0.26) | -0.53 (0.44)
  the refractive error 1 month postoperative | -0.37 (0.24) | -0.46 (0.47)
  the refractive error 3 month postoperative | -0.36 (0.23) | -0.48 (0.22)
  the refractive error 6 months postoperative | -0.41 (0.22) | -0.48 (0.21)

ADVERSE EVENTS:
Arm/Group | Cataract
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes